CLINICAL TRIAL: NCT06227598
Title: From Nature to Bedside- Algae Based Bio Compound for Prevention and Treatment of Inflammation, Pain and IBD
Acronym: Algae4IBD
Status: Not yet recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Felice Amato, Associate Professor, Federico II University
Other Study IDs: ALGAE4IBD
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Procedure: Additional biopsies collection — Procedure: Additional biopsies collection We will recruit only subjects (UC, CD and NO-UC/CD) scheduled for the endoscopy and biopsies-collection according to the usual clinical practice. During the endoscopy we will collect 6 additional biopsies.

SUMMARY:
This study is part of the project funded by the Horizon2020 program for establishing the consortium Algae4IBD (https://algae4ibd.eu/), where Dept. of Molecular Medicine and Medical Biotechnologies (DMMBM) University of Naples Federico II participates as a partner. It aims to promote the implementation of the European Crohn's and Colitis Organization (ECCO/FECCO) Directive and the benefit of the Inflammatory Bowel Disease (IBD) patient's wellness by finding innovative algae based novel small molecule therapeutics. A systemic approach to eco-innovation is adopted to create interconnections between sectors, value chains, natural resources, and relevant societal stewards. To this end, the consortium has set specific objectives to achieve holistic innovations, including technical, economic, health, and social factors that all work in concert.

IBD included Crohn's disease and ulcerative colitis. It is a class of chronic inflammatory disorders with complex pathogenesis. Despite the lack of a full understanding of its etiogenesis, many anti-inflammatory treatments have been developed over the last decades. However, not all patients may benefit from these treatments and some of them are refractory to the current therapies or experience relapse of the disease. Therefore, there is still an urgent need to find an innovative line of interventions for ameliorating these patients' overall quality of life.

Algae4IBD consortium will form a bridge between innovation and market demands to prevent and treat inflammation, pain, and IBD. Bioactive molecule/compounds extracts from microalgae, cyanobacteria, and macro-algae (MiaCyMa) are an inexhaustible untapped natural source for products destined for IBD prevention and treatment (inflammation, pain, and the disease process associated with the gut's microbiome). The natural source potential is still more promising when considering extremophile strains for excellent metabolism systems. Moreover, the production of the natural source of biological materials should be sustainable. Indeed, the non-genetically modified organisms (GMO cultures offer numerous advantages such as reduced requirements of fresh water and land (no arable land is required), drastic reduction of nitrogen sources, and potential environmental threats. Algae4IBD concept will include a multi-step screening approach and feedback loops across the project steps to achieve its goals. Specifically, DMMBM is in charge with work package (WP) 4, task 4.4.2, which aims to characterize the activity of plant cell (algae) extracts named in this proposal as "natural compounds" of algae provided by the consortium in ex-vivo models, using bioptic samples derived from patients with IBD (patients with ulcerative colitis (UC) and Crohn's disease (CD)), comparing them to samples derived from patients without UC and CD.

ELIGIBILITY:
Inclusion Criteria:

SUBJECTS WITH THE DIAGNOSIS OF UC OR CD:

* subjects undergoing endoscopy and biopsies collection per standard of care
* patients ≥2 and <60 years

Additionally, for people with UC:

- clinical and endoscopic evaluation (Mayo score≥2)

Additionally, for individuals with CD:

- clinical and endoscopic evaluation (Harvey-Bradshaw score ≥5 and overall simplified endoscopic score (SES-CD) >2)

SUBJECTS NOT AFFECTED BY UC OR CD:

subjects undergoing endoscopy and biopsies collection (≥2 and <60 years) according to the normal clinical practice (as patients undergoing cancer surveillance, irritable bowel syndrome (IBS), diarrhea) subjects not affected by UC or CD according to the previously reported clinical and endoscopic evaluation criteria All patients will sign the informed consent.

Exclusion Criteria:

SUBJECTS WITH THE DIAGNOSIS OF UC OR CD:

- subjects with UC or CD who do not have the previously described clinical and endoscopic evaluation criteria

SUBJECTS NOT AFFECTED BY UC OR CD (CONTROL GROUP):

-subjects undergoing anti-inflammatory and/or immunosuppressive treatments for other diseases not related to UC or CD

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * : Ulcerative Colitis (UC)
    1. subjects undergoing endoscopy and biopsies collection per standard of care
    2. adult patients ≥2 and <60 years
    3. clinical and endoscopic evaluation (Mayo score≥2)
  * : Crohn's Disease (CD)
    1. subjects undergoing endoscopy and biopsies collection per standard of care
    2. adult patients ≥2 and <60 years
    3. clinical and endoscopic evaluation (Harvey-Bradshaw score ≥5 and overall simplified endoscopic score (SES-CD) >2)
  * : NO UC/CD
    1. subjects undergoing endoscopy and biopsies collection (≥2 and <60 years) according to the normal clinical practice (as patients undergoing cancer surveillance, irritable bowel syndrome (IBS), diarrhea)
    2. subjects not affected by UC or CD according to the previously reported clinical and endoscopic evaluation criteria
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the response of intestinal mucosa samples to treatments with natural compounds derived from algae in terms of release of pro-inflammatory factors (1), and epithelium barrier integrity (2) | 30 months
  1. Release of pro-inflammatory cytokines using ELISA
  2. Epithelium integrity measurement through transepithelial electrical resistance (TEER) evaluation and Ussing chamber analysis.
  By multi-assay factor analysis we will integrate these data with the patients' clinical parameters, correlating among each other in parallel and giving one single output (outcome measure, in our case) explaining how the different data are assigned simultaneously to specific clinical characteristics, thus resulting as associated with, or predictive of, the clinical progression of IBD

IPD SHARING:
Plan to Share IPD: Undecided